CLINICAL TRIAL: NCT03916042
Title: A Multi-Center, Phase 2, Randomized, Double-Masked, Parallel-Group, Vehicle-Controlled, Clinical Trial to Assess the Safety and Efficacy of Reproxalap Ophthalmic Solution (0.25% Novel Formulation) Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: A Multi-Center, Randomized, Double-Masked, Parallel-Group, Vehicle-Controlled, Clinical Trial of Reproxalap to Assess the Safety and Efficacy in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-DED-013
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2023-02

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reproxalap (0.25% Novel Formulation) QID to BID (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25% Novel Formulation) QID to BID
- Vehicle Ophthalmic Solution QID to BID (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution (0.25% Novel Formulation) QID to BID

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25% Novel Formulation) QID to BID — Reproxalap Opthalmic Solution (0.25% Novel Formulation) administered QID for four weeks, followed by BID administration for eight weeks
  Arms: Reproxalap (0.25% Novel Formulation) QID to BID
Drug: Vehicle Ophthalmic Solution (0.25% Novel Formulation) QID to BID — Vehicle Ophthalmic Solution administered QID for four weeks, followed by BID administration for eight weeks
  Arms: Vehicle Ophthalmic Solution QID to BID

SUMMARY:
A Multi-Center, Phase 2, Randomized, Double-Masked, Parallel-Group, Vehicle-Controlled, Clinical Trial to Assess the Safety and Efficacy of Reproxalap Ophthalmic Solution (0.25% Novel Formulation) Compared to Vehicle in Subjects with Dry Eye Disease

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age of either gender and any race;
* Have a reported history of dry eye for at least 6 months prior to Visit 1;
* Have a history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1

Exclusion Criteria:

* Have any clinically significant slit-lamp findings at Visit 1, including active blepharitis; meibomian gland dysfunction (MGD); lid margin inflammation; or active ocular allergies that require therapeutic treatment, or, in the opinion of the investigator may interfere with the assessment of the safety or efficacy of reproxalap or vehicle;
* Have or be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal) or active ocular inflammation at Visit 1;
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
* Have used any eye drops within 2 hours of Visit 1;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Have used ophthalmic cyclosporine or lifitegrast 5.0% ophthalmic solution within 90 days of Visit 1;
* Have any planned ocular and/or lid surgeries over the study period or any ocular surgery within 6 months of Visit 1;
* Have used temporary or permanent punctal plugs within 30 days prior to Visit 1 or anticipate their use during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Reproxalap (0.25% Novel Formulation): Reproxalap ophthalmic solution administered QID (four times daily) for four weeks, followed by BID (two times daily) administration for eight weeks
- Vehicle: Vehicle ophthalmic solution administered QID for four weeks, followed by BID administration for eight weeks
Period: Overall Study
Arm/Group | Reproxalap (0.25% Novel Formulation) | Vehicle
Started | 102 | 104
Completed | 96 | 97
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Reproxalap (0.25% Novel Formulation): Reproxalap ophthalmic solution administered QID for four weeks, followed by BID administration for eight weeks
- Total: Total of all reporting groups
Arm/Group | Reproxalap (0.25% Novel Formulation) | Vehicle | Total
Number analyzed (Participants) | 102 | 104 | 206
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 58 | 110
  >=65 years | 50 | 46 | 96
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 69 | 151
  Male | 20 | 35 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 94 | 96 | 190
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 5 | 6
  Black or African American | 10 | 14 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 89 | 83 | 172
  Multiple | 0 | 1 | 1
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 102 | 104 | 206
Iris Color (Right Eye) [Count of Participants; unit: Participants]
  Black | 0 | 3 | 3
  Blue | 28 | 27 | 55
  Brown | 46 | 44 | 90
  Hazel | 21 | 20 | 41
  Gray | 1 | 1 | 2
  Green | 6 | 9 | 15
  Other | 0 | 0 | 0
Iris Color (Left Eye) [Count of Participants; unit: Participants]
  Black | 0 | 3 | 3
  Blue | 28 | 27 | 55
  Brown | 46 | 44 | 90
  Hazel | 21 | 20 | 41
  Gray | 1 | 1 | 2
  Green | 6 | 9 | 15
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Subject-reported Ocular Dryness Score (0 - 100 Visual Analogue Scale (VAS))
Description: Change from baseline comparison of reproxalap to vehicle for subject-reported Ocular Dryness Score VAS (0 = no discomfort - 100 = maximal discomfort), where a higher score means a worse outcome. The intervention was administered bilaterally. The Least Squares Mean (standard error) was derived from mixed model repeated measures for change from baseline calculated using baseline score, treatment arm, visit, and the interaction of treatment arm and visit as fixed effects.
Time Frame: Efficacy assessment period (Day 1 through 85) - assessed at Weeks 1, 2, 4, 6, 8, 10, and 12. Baseline was Day 1.
Population: Intent-to-treat Ocular Dryness Population with observed data only
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Reproxalap (0.25% Novel Formulation) | Vehicle
Number analyzed (Participants) | 82 | 83
score on a scale | -16.0 (2.20) | -9.1 (2.18)

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected for each subject in the clinical trial was approximately three months.
Arm/Group | Reproxalap (0.25% Novel Formulation) | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/104
Serious Adverse Events (participants affected / at risk) | 1/102 | 1/104
Other Adverse Events (participants affected / at risk) | 91/102 | 8/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap (0.25% Novel Formulation) (N=102) | Vehicle (N=104)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 — The serious adverse event of cellulitis was deemed moderate in severity and not related to study drug by the Principal Investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap (0.25% Novel Formulation) (N=102) | Vehicle (N=104)
Visual acuity reduced (Eye disorders) | 9 | 4 — All visual acuity reduced adverse events were deemed mild in severity by the Principal Investigators.
General disorders and administration site conditions (General disorders) | 82 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT03916042/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT03916042/SAP_001.pdf